CLINICAL TRIAL: NCT06641206
Title: Intra-articular Dexmedetomidine for Treatment of Chronic Knee Pain: A Prospective Case-Control Clinical Trial
Brief Title: Intra-Articular Dexmedetomidine: A Treatment for Chronic Knee Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed ElKashef, lecturer of Anesthesia and Surgical ICU, Faculty of Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR843/9/24
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Knee Pain
MeSH Terms: interventions — Triamcinolone Acetonide; Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): A group of Patients from Tanta University suffering from Chronic painful knee osteoarthritis who didn't receive medical treatment and progressed to have chronic pain with decreased physical function and poorer quality of life.
  Interventions: Drug: Triamcinolone Acetonide; Drug: Bupivacaine Hydrochloride
- Group 2 (Active Comparator): A group of Patients from Tanta University suffering from Chronic painful knee osteoarthritis who didn't receive medical treatment and progressed to have chronic pain with decreased physical function and poorer quality of life.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Triamcinolone Acetonide — 1 ml of triamcinolone acetonide was used to prepare a solution for knee injection for patients with Chronic Knee Pain
  Arms: Group 1
Drug: Bupivacaine Hydrochloride — 20mg of bupivacaine hydrochloride was used to prepare a solution for knee injection for patients with Chronic Knee Pain
  Arms: Group 1
Drug: Dexmedetomidine — Dexmedetomidine solution was prepared by mixing Dexmedetomidine in a dose of 3 µg/kg in 5-ml saline
  Arms: Group 2

SUMMARY:
Chronic knee osteoarthritis (KOA) is a painful condition with limited treatment options. Non-pharmacological approaches often fall short, leading to decreased quality of life. Ozone therapy, a simple and affordable treatment, has shown promise for pain relief. Dexmedetomidine (DEX), a sedative and analgesic, has been used successfully as an adjuvant to anesthesia and local anesthetics. Given its potential for pain management, exploring DEX as a treatment for KOA could offer a new and promising approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients were not assigned for surgical intervention;
* Patients were free of exclusion criteria

Exclusion Criteria:

* Patients were assigned for surgical intervention;
* Patients who had uncontrolled hypertension and/or diabetes mellitus;
* Patients who had uncompensated cardiac, renal, or hepatic diseases;
* Patients with coagulopathy, spinal deformity, allergy, or contraindication for the used drugs;
* Patients who refused to sign the informed consent were excluded from the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% reduction in pain (measured by Numerical Rating Scale) post-intra-articular Injection. | 7 months
  Value of intra-articular Injection in Pain Reduction of chronic knee pain manifested by recurrence of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbyia, Egypt